CLINICAL TRIAL: NCT03136380
Title: A Single Centre, Double Blind (Sponsor Open), Placebo Controlled, 3-Period Crossover, Ascending Dose Study in Japanese Healthy Elderly Male Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of Danirixin in the Fed State (Part1) and an Open Label, 2-way Crossover to Evaluate Food Effect on the Pharmacokinetics of Danirixin (Part2)
Brief Title: Study of Danirixin in Japanese Healthy Elderly Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 206817
Record Dates: First submitted 2017-04-17; First posted 2017-05-02 (Actual); Results first posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: healthy Japanese subjects; CXCR2 inhibitor; Danirixin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1: Group A (Experimental): Subjects will receive GSK1325756H 10 mg in P-1, GSK1325756H 50 mg in P-2 and placebo in P-3 after a high fat meal. There will be a washout period of at least 7 days between each treatment period.
  Interventions: Drug: GSK1325756H; Drug: Placebo
- Part 1: Group B (Experimental): Subjects will receive GSK1325756H 10 mg in P-1, placebo in P-2 and GSK1325756H 100 mg in P-3 after a high fat meal. There will be a washout period of at least 7 days between each treatment period.
  Interventions: Drug: GSK1325756H; Drug: Placebo
- Part 1: Group C (Experimental): Subjects will receive placebo in P-1, GSK1325756H 50 mg in P-2 and GSK1325756H 100 mg in P-3 after a high fat meal. There will be a washout period of at least 7 days between each treatment period.
  Interventions: Drug: GSK1325756H; Drug: Placebo
- Part 2: Group D (Experimental): Subjects will receive GSK1325756H 50 mg after a low fat meal and fasted state respectively. There will be a washout period of at least 7 days between each treatment period.
  Interventions: Drug: GSK1325756H
- Part 2: Group E (Experimental): Subjects will receive GSK1325756H 50 mg after a fasted state and a low fat meal respectively. There will be a washout period of at least 7 days between each treatment period.
  Interventions: Drug: GSK1325756H

INTERVENTIONS:
Drug: GSK1325756H — Danirixin will be available as 10 and 50 milligram (mg) white film coated, round and oval tablets intended for oral administration. It will be administered with 240 mL of water.
Drug: Placebo — Subjects will receive visually matching danirixin placebo tablets. It will be administered with 240 mL of water.
  Arms: Part 1: Group A; Part 1: Group B; Part 1: Group C

SUMMARY:
Danirixin is a selective chemokine receptor antagonist being developed as a potential anti-inflammatory agent for the treatment of chronic obstructive pulmonary disease (COPD). The aim of the study is to assess the safety, tolerability and pharmacokinetics (PK) in healthy Japanese subjects over the age of 65 years (inclusive). The study will be conducted in two parts: Part 1 will be a double blind, placebo-controlled, 3-period crossover, ascending single oral dose administration of GSK1325756H (Hydrobromide Salt Tablet Formulations of Danirixin) 10, 50 and 100 milligram (mg) in the fed condition. Part 2 will be an open label, 2-period crossover, single oral dose of GSK1325756H 50 mg in fed and fasted state. This study will provide an understanding of PK of hydrobromide salt of GSK1325756 in population of healthy elderly subjects and also contribute to the selection of appropriate dosing for Phase IIa study in Japan.

ELIGIBILITY:
Inclusion Criteria

* Participant must be over 65 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECG. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Participants whose peripheral blood neutrophil counts and hematocrit values are within normal range at screening visit.
* Body weight >=50 kilogram (Kg) and body mass index (BMI) within the range 18.5-24.9 kg/square meter (m^2) (inclusive).
* Japanese Male: A male participant must agree to use contraception during the treatment period and until follow up visit.
* Capable of giving signed informed consent.

Exclusion Criteria

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Abnormal blood pressure as determined by the investigator.
* Alanine Aminotransferase (ALT)>1.5x upper limit of normal (ULN).
* Bilirubin>1.5xULN (isolated bilirubin > 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF)> 450 millisecond (msec).
* Past or intended use of over-the-counter or prescription medication including herbal medications and proton pump inhibitor (PPI) within 14 days prior to dosing.
* History of donation of blood or blood products >=400 milliliter (mL) within 3 months or >=200 mL within 1 month prior to screening.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation within the last 30 days before signing of consent in this clinical study involving an investigational study treatment or any other type of medical research.
* The subject with positive Serological test for syphilis (Rapid Plasma Reagin [RPR] and Treponema pallidum hemagglutination test [TPHA]), Human immunodeficiency virus (HIV) Antigen/Antibody, Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody, or Human T-cell lymphotropic virus type 1 (HTLV-1) antibody at screening.
* Positive pre-study drug screen.
* Regular alcohol consumption within 6 months prior to the study defined as: an average weekly intake of > 14 units for males. One unit is equivalent to 350 mL of beer, 150 mL of wine or 45 mL of 80 proof distilled spirits.
* Smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Japanese Healthy Elderly Male Subjects
Enrollment: 34 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Tokyo, Japan

REFERENCES:
- [Derived] Iida T, Matsuzawa Y, Ogura H, Nagakubo T, Wakamatsu A, Ambery C, Miller BE, Lazaar AL, Numachi Y. Evaluation of the Safety, Tolerability, Pharmacokinetics, and Food Effect of Danirixin Hydrobromide Tablets in Japanese Healthy Elderly Participants. Clin Pharmacol Drug Dev. 2019 Nov;8(8):1081-1087. doi: 10.1002/cpdd.693. Epub 2019 May 6. PMID 31056840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in Tokyo, Japan from 10-May-2017 to 31-July-2017.
Pre-assignment Details: A total of 147 participants were screened of which 113 were screen failures the reasons of which were investigator discretion (1), lost to follow-up (2) screened but enrollment target reached prior to enrollment (5) and did not met inclusion/exclusion criteria (105). A total of 18 participants in Part 1 and 16 in Part 2 were enrolled in the study.
Groups:
- Part 1-GSK1325756H 10 mg Then GSK1325756H 50 mg Then Placebo: Participants in this arm received GSK1325756H 10 milligrams (mg) in treatment period 1 followed by GSK1325756H 50 mg in treatment period 2 followed by placebo in treatment period 3. The treatment periods were separated were separated by a minimum of one-week washout period.
- Part 1-GSK1325756H 10 mg Then Placebo Then GSK1325756H 100 mg: Participants in this arm received GSK1325756H 10 mg in treatment period 1 followed placebo in treatment period 2 followed by GSK1325756H 100 mg in treatment period 3. The treatment periods were separated were separated by a minimum of one-week washout period.
- Part 1-Placebo Then GSK1325756H 50 mg Then GSK1325756H 100 mg: Participants in this arm received placebo in treatment period 1 followed by GSK1325756H 50 mg in treatment period 2 followed by GSK1325756H 100 mg in treatment period 3. The treatment periods were separated were separated by a minimum of one-week washout period.
- Part 2-GSK1325756H Fed Followed by Fasted: Participants were randomized to receive GSK1325756H 50 mg (fed) in Period 1 followed by GSK1325756H (fasted) in Period 2 of Part 2. The treatment periods were separated were separated by a minimum of one-week washout period.
- Part 2-GSK1325756H Fasted Followed by Fed: Participants were randomized to receive GSK1325756H 50 mg (fasted) in Period 1 followed by GSK1325756H (fed) in Period 2 of Part 2. The treatment periods were separated were separated by a minimum of one-week washout period.
Period: Part 1, Period 1 (3 Days)
Arm/Group | Part 1-GSK1325756H 10 mg Then GSK1325756H 50 mg Then Placebo | Part 1-GSK1325756H 10 mg Then Placebo Then GSK1325756H 100 mg | Part 1-Placebo Then GSK1325756H 50 mg Then GSK1325756H 100 mg | Part 2-GSK1325756H Fed Followed by Fasted | Part 2-GSK1325756H Fasted Followed by Fed
Started | 6 | 6 | 6 | 0 | 0
Completed | 6 | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 1, Washout Period 1 (7 Days)
Arm/Group | Part 1-GSK1325756H 10 mg Then GSK1325756H 50 mg Then Placebo | Part 1-GSK1325756H 10 mg Then Placebo Then GSK1325756H 100 mg | Part 1-Placebo Then GSK1325756H 50 mg Then GSK1325756H 100 mg | Part 2-GSK1325756H Fed Followed by Fasted | Part 2-GSK1325756H Fasted Followed by Fed
Started | 6 | 6 | 6 | 0 | 0
Completed | 6 | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 1, Period 2 (3 Days)
Arm/Group | Part 1-GSK1325756H 10 mg Then GSK1325756H 50 mg Then Placebo | Part 1-GSK1325756H 10 mg Then Placebo Then GSK1325756H 100 mg | Part 1-Placebo Then GSK1325756H 50 mg Then GSK1325756H 100 mg | Part 2-GSK1325756H Fed Followed by Fasted | Part 2-GSK1325756H Fasted Followed by Fed
Started | 6 | 6 | 6 | 0 | 0
Completed | 6 | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 1, Washout Period 2 (7 Days)
Arm/Group | Part 1-GSK1325756H 10 mg Then GSK1325756H 50 mg Then Placebo | Part 1-GSK1325756H 10 mg Then Placebo Then GSK1325756H 100 mg | Part 1-Placebo Then GSK1325756H 50 mg Then GSK1325756H 100 mg | Part 2-GSK1325756H Fed Followed by Fasted | Part 2-GSK1325756H Fasted Followed by Fed
Started | 6 | 6 | 6 | 0 | 0
Completed | 6 | 5 | 6 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Period: Part 1, Period 3 (4 Days)
Arm/Group | Part 1-GSK1325756H 10 mg Then GSK1325756H 50 mg Then Placebo | Part 1-GSK1325756H 10 mg Then Placebo Then GSK1325756H 100 mg | Part 1-Placebo Then GSK1325756H 50 mg Then GSK1325756H 100 mg | Part 2-GSK1325756H Fed Followed by Fasted | Part 2-GSK1325756H Fasted Followed by Fed
Started | 6 | 5 | 6 | 0 | 0
Completed | 6 | 5 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2, Period 1 (3 Days)
Arm/Group | Part 1-GSK1325756H 10 mg Then GSK1325756H 50 mg Then Placebo | Part 1-GSK1325756H 10 mg Then Placebo Then GSK1325756H 100 mg | Part 1-Placebo Then GSK1325756H 50 mg Then GSK1325756H 100 mg | Part 2-GSK1325756H Fed Followed by Fasted | Part 2-GSK1325756H Fasted Followed by Fed
Started | 0 | 0 | 0 | 8 | 8
Completed | 0 | 0 | 0 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2, Washout Period 1 (7 Days)
Arm/Group | Part 1-GSK1325756H 10 mg Then GSK1325756H 50 mg Then Placebo | Part 1-GSK1325756H 10 mg Then Placebo Then GSK1325756H 100 mg | Part 1-Placebo Then GSK1325756H 50 mg Then GSK1325756H 100 mg | Part 2-GSK1325756H Fed Followed by Fasted | Part 2-GSK1325756H Fasted Followed by Fed
Started | 0 | 0 | 0 | 8 | 8
Completed | 0 | 0 | 0 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2, Period 2 (3 Days)
Arm/Group | Part 1-GSK1325756H 10 mg Then GSK1325756H 50 mg Then Placebo | Part 1-GSK1325756H 10 mg Then Placebo Then GSK1325756H 100 mg | Part 1-Placebo Then GSK1325756H 50 mg Then GSK1325756H 100 mg | Part 2-GSK1325756H Fed Followed by Fasted | Part 2-GSK1325756H Fasted Followed by Fed
Started | 0 | 0 | 0 | 8 | 8
Completed | 0 | 0 | 0 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1-Total Participants: Participants received a single dose of GSK1325756H 10 mg (fed), GSK1325756 50 mg (fed), GSK1325756 100 mg (fed) and matching placebo in one of the three treatment periods in a crossover manner. The treatment periods were separated by a minimum of one-week washout period. The maximum duration of participation of participants, in Part 1 was 24 days.
- Part 2-Total Participants: Participants received a single dose of GSK1325756 50 mg (fed) and GSK1325756 50 mg (fasted) in one of the two treatment periods in a crossover manner. The treatment periods were separated by a minimum of one-week washout period. The maximum duration of participation of participants, in Part 2 was 13 days.
- Total: Total of all reporting groups
Arm/Group | Part 1-Total Participants | Part 2-Total Participants | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.0 (3.01) | 69.3 (2.89) | 69.6 (2.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 16 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese/East Asian /South East Asian Heritage | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) and Serious Adverse Events in Part 1
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. Safety population comprised of all participants who took at least one dose of study treatment.
Time Frame: Up to 32 days in Part 1
Population: Safety Population
Measure: Number; unit: Participants
Groups:
- Part 1: Placebo (Fed): Participants received matching placebo tablets via the oral route with food (fed state) and 240 milliliters of water in Part 1.
- Part 1: GSK1325756H 10 mg (Fed): Participants received GSK1325756H 10 mg tablets via the oral route with food (fed state) and 240 milliliters of water in Part 1.
- Part 1: GSK1325756H 50 mg (Fed): Participants received GSK1325756H 50 mg tablets via the oral route with food (fed state) and 240 milliliters of water in Part 1.
- Part 1: GSK1325756H 100 mg (Fed): Participants received GSK1325756H 100 mg tablets via the oral route with food (fed state) and 240 milliliters of water in Part 1.
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Participants
  Any AE | 1 | 0 | 0 | 1
  Any SAE | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Any Adverse Event (AE) and Serious Adverse Events in Part 2
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant
Time Frame: Up to 21 days in Part 2
Population: Safety Population
Measure: Number; unit: Participants
Groups:
- Part 2: GSK1325756H 50 mg (Fed): Participants received GSK1325756H 50 mg tablets via the oral route with food (fed state) and 240 milliliters of water in Part 2.
- Part 2: GSK1325756H 50 mg (Fasted): Participants received GSK1325756H 50 mg tablets via the oral route without food (fasted state) and 240 milliliters of water in Part 2.
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Participants
  Any AE | 1 | 0
  Any SAE | 0 | 0

3. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters Calcium, Cholesterol, Chloride, Glucose, High Density Lipids (HDL) Cholesterol, Potassium, Low Density Lipids (LDL) Cholesterol,Sodium,Phosphorus,Triglycerides,Urea/Blood Urea Nitrogen (BUN) in Part 1
Description: Blood samples were collected for the assessment of chemistry parameters namely calcium, cholesterol, chloride, glucose, HDL cholesterol, potassium, LDL cholesterol, sodium, phosphorus, triglycerides, and urea/BUN results for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles/liter
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Millimoles/liter
  Calcium, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Calcium, 48 hours | -0.0208 (0.04617) | -0.0187 (0.04137) | 0.0021 (0.05675) |
  Calcium, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Calcium, 72 hours | -0.0000 (0.06312) |  |  | -0.0318 (0.05124)
  Cholesterol, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Cholesterol, 48 hours | 0.0453 (0.36206) | 0.0129 (0.30588) | 0.1681 (0.53220) |
  Cholesterol, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Cholesterol, 72 hours | 0.2241 (0.62379) |  |  | -0.0541 (0.37997)
  Chloride, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Chloride, 48 hours | 1.8 (1.11) | 1.9 (1.83) | 1.9 (1.44) |
  Chloride, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Chloride, 72 hours | 1.8 (1.17) |  |  | 1.5 (1.75)
  Glucose, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Glucose, 48 hours | 0.2452 (0.27852) | 0.3516 (0.34246) | 0.1619 (0.32580) |
  Glucose, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Glucose, 72 hours | 0.2776 (0.16088) |  |  | 0.1463 (0.38958)
  HDL cholesterol, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  HDL cholesterol, 48 hours | -0.1789 (0.16035) | -0.1702 (0.12302) | -0.1228 (0.13910) |
  HDL cholesterol, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  HDL cholesterol, 72 hours | -0.1509 (0.11380) |  |  | -0.2304 (0.10753)
  Potassium, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Potassium, 48 hours | 0.04 (0.162) | 0.11 (0.231) | 0.28 (0.359) |
  Potassium, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Potassium, 72 hours | -0.17 (0.294) |  |  | 0.07 (0.200)
  LDL cholesterol, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  LDL cholesterol, 48 hours | -0.0065 (0.35150) | 0.0043 (0.26961) | 0.0711 (0.44012) |
  LDL cholesterol, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  LDL cholesterol, 72 hours | 0.1896 (0.56007) |  |  | -0.0188 (0.36555)
  Sodium, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Sodium, 48 hours | 0.6 (1.00) | 1.4 (2.07) | 0.9 (1.08) |
  Sodium, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Sodium, 72 hours | 1.0 (0.89) |  |  | 1.1 (1.45)
  Phosphorus, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Phosphorus, 48 hours | -0.1588 (0.12039) | -0.1399 (0.08525) | -0.1426 (0.09972) |
  Phosphorus, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Phosphorus, 72 hours | -0.0969 (0.05776) |  |  | -0.1262 (0.11041)
  Triglycerides, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Triglycerides, 48 hours | 0.6422 (0.31917) | 0.4963 (0.36405) | 0.5575 (0.38005) |
  Triglycerides, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Triglycerides, 72 hours | 0.3823 (0.34016) |  |  | 0.4910 (0.21744)
  Urea/BUN, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Urea/BUN, 48 hours | -0.7140 (0.79099) | -0.5355 (1.14422) | -0.1785 (0.95672) |
  Urea/BUN, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Urea/BUN, 72 hours | -0.2975 (0.41735) |  |  | -0.5193 (0.96276)

4. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters Alkaline Phosphatase, Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Creatine Kinase, Gamma Glutamyl Transferase (GGT) and Lactate Dehydrogenase for Part 1
Description: Blood samples were collected for the assessment of chemistry parameters namely alkaline phosphatase, ALT, AST, creatine kinase, GGT and lactate dehydrogenase for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units/liter
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
International units/liter
  Alkaline phosphatase, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Alkaline phosphatase, 48 hours | 1.1 (9.08) | -1.5 (8.44) | 0.0 (9.55) |
  Alkaline phosphatase,72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Alkaline phosphatase,72 hours | 12.5 (13.37) |  |  | 4.6 (12.14)
  ALT, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  ALT, 48 hours | -2.2 (2.89) | -0.5 (3.92) | -1.9 (2.94) |
  ALT, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  ALT, 72 hours | 2.5 (3.83) |  |  | 0.6 (2.29)
  AST, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  AST, 48 hours | -2.3 (4.38) | -0.6 (4.52) | -2.2 (3.19) |
  AST, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  AST, 72 hours | 1.5 (3.67) |  |  | -1.4 (2.11)
  Creatine kinase, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Creatine kinase, 48 hours | -29.0 (27.10) | -34.3 (23.83) | -32.3 (22.18) |
  Creatine kinase, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Creatine kinase, 72 hours | -34.7 (9.99) |  |  | -46.4 (32.96)
  GGT, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  GGT, 48 hours | -1.0 (1.48) | 0.9 (1.44) | -1.9 (2.35) |
  GGT, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  GGT, 72 hours | 2.0 (1.10) |  |  | -0.1 (1.70)
  Lactate dehydrogenase, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Lactate dehydrogenase, 48 hours | -15.3 (20.20) | -13.8 (11.66) | -12.0 (10.08) |
  Lactate dehydrogenase, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Lactate dehydrogenase, 72 hours | -2.8 (49.15) |  |  | -17.3 (7.40)

5. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters Albumin and Total Protein for Part 1
Description: Blood samples were collected for the assessment of chemistry parameters namely albumin and total protein for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams/liter
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Grams/liter
  Albumin, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Albumin, 48 hours | -0.3 (1.44) | -0.6 (1.44) | 0.3 (1.96) |
  Albumin, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Albumin, 72 hours | 1.2 (2.32) |  |  | -1.0 (1.34)
  Total protein, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Total protein, 48 hours | 0.2 (2.59) | -0.3 (1.82) | 0.8 (3.01) |
  Total protein, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Total protein, 72 hours | 1.8 (2.64) |  |  | 0.0 (2.49)

6. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid for Part 1
Description: Blood samples were collected for the assessment of chemistry parameters namely direct bilirubin, total bilirubin, creatinine and uric acid for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles/liter
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Micromoles/liter
  Direct bilirubin, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Direct bilirubin, 48 hours | -0.428 (0.7734) | 0.000 (1.2629) | -0.712 (0.8805) |
  Direct bilirubin, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Direct bilirubin, 72 hours | -0.855 (1.4307) |  |  | -0.466 (0.7987)
  Total bilirubin, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Total bilirubin, 48 hours | -1.283 (2.0784) | -0.428 (3.3513) | -1.425 (1.9060) |
  Total bilirubin, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Total bilirubin, 72 hours | -2.565 (4.6830) |  |  | -2.332 (1.7560)
  Creatinine, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Creatinine, 48 hours | -1.9890 (4.33275) | -3.6833 (3.21689) | -1.8417 (3.02629) |
  Creatinine, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Creatinine, 72 hours | -4.7147 (3.73658) |  |  | -4.0985 (3.79755)
  Uric acid, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Uric acid, 48 hours | -33.7053 (25.78160) | -33.7053 (17.26380) | -31.7227 (21.57043) |
  Uric acid, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Uric acid, 72 hours | -27.7573 (43.97767) |  |  | -23.2513 (23.10621)

7. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter Amylase for Part 1
Description: Blood samples were collected for the assessment of chemistry parameters namely amylase for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Units/liter
  Amylase, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Amylase, 48 hours | 16.0 (9.16) | 20.6 (18.05) | 22.7 (13.21) |
  Amylase, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Amylase, 72 hours | 38.8 (28.84) |  |  | 14.4 (12.92)

8. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters Calcium, Cholesterol, Chloride, Glucose, HDL Cholesterol, Potassium, LDL Cholesterol, Sodium, Phosphorus Inorganic, Triglycerides, Urea/BUN for Part 2
Description: Blood samples were collected for the assessment of chemistry parameters namely calcium, cholesterol, chloride, glucose, HDL cholesterol, potassium, LDL cholesterol, sodium, phosphorus, triglycerides, urea/BUN results for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles/liter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Millimoles/liter
  Calcium, 48 hours | 0.0000 (0.05834) | 0.0000 (0.05154)
  Cholesterol, 48 hours | 0.3119 (0.37218) | 0.3588 (0.25265)
  Chloride, 48 hours | 0.2 (2.01) | 0.5 (1.86)
  Glucose, 48 hours | 0.2116 (0.23744) | 0.1561 (0.35643)
  HDL cholesterol, 48 hours | -0.1131 (0.12629) | -0.0808 (0.10678)
  Potassium, 48 hours | 0.18 (0.377) | 0.14 (0.326)
  LDL cholesterol, 48 hours | 0.1729 (0.30124) | 0.2279 (0.27614)
  Sodium, 48 hours | -0.3 (1.65) | 0.8 (1.72)
  Phosphorus inorganic, 48 hours | -0.0868 (0.08561) | -0.1433 (0.08821)
  Triglycerides, 48 hours | 0.7402 (0.43390) | 0.6010 (0.39556)
  Urea/BUN, 48 hours | -0.6024 (1.44409) | -0.3347 (0.90755)

9. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters Alkaline Phosphatase, ALT, AST, Creatine Kinase, GGT and Lactate Dehydrogenase for Part 2
Description: Blood samples were collected for the assessment of chemistry parameters namely alkaline phosphatase, ALT, AST, creatine kinase, GGT and lactate dehydrogenase for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units/liter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
International units/liter
  Alkaline phosphatase, 48 hours | 0.9 (9.96) | 6.5 (11.35)
  ALT, 48 hours | -1.5 (1.93) | -1.5 (1.97)
  AST, 48 hours | -2.0 (2.28) | -1.8 (1.29)
  Creatine kinase, 48 hours | -29.7 (28.72) | -16.6 (18.89)
  GGT, 48 hours | -0.5 (2.99) | -0.4 (2.50)
  Lactate dehydrogenase, 48 hours | -14.8 (11.97) | -13.7 (6.80)

10. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters Albumin and Total Protein for Part 2
Description: Blood samples were collected for the assessment of chemistry parameters namely albumin and total protein for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams/liter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Grams/liter
  Albumin, 48 hours | 0.3 (1.54) | 0.8 (1.48)
  Total protein, 48 hours | 1.1 (2.66) | 1.9 (2.25)

11. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid for Part 2
Description: Blood samples were collected for the assessment of chemistry parameters namely direct bilirubin, total bilirubin, creatinine and uric acid for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles/liter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Micromoles/liter
  Direct bilirubin, 48 hours | -0.641 (1.5135) | -0.641 (1.2291)
  Total bilirubin, 48 hours | -1.496 (4.6254) | -0.748 (2.6468)
  Creatinine, 48 hours | -2.8178 (3.68348) | -4.2542 (3.32677)
  Uric acid, 48 hours | -15.6135 (54.03085) | -8.5502 (75.89141)

12. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter Amylase for Part 2
Description: Blood samples were collected for the assessment of chemistry parameter namely amylase for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Units/liter | 18.2 (8.63) | 18.5 (8.75)

13. Primary Outcome: Change From Baseline in Hematology Parameters Basophils, Eosinophils, Lymphocytes, Monocytes and Total Neutrophils for Part 1
Description: Blood samples were collected for the assessment of hematology parameters namely basophils, eosinophils, leukocytes, lymphocytes, monocytes, total neutrophils and platelets for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Percentage of cells
  Basophils, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Basophils, 48 hours | 0.12 (0.221) | 0.09 (0.168) | 0.09 (0.131) |
  Basophils, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Basophils, 72 hours | 0.13 (0.082) |  |  | 0.03 (0.272)
  Eosinophils, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Eosinophils, 48 hours | 1.39 (1.132) | 0.95 (1.301) | 0.73 (0.725) |
  Eosinophils, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Eosinophils, 72 hours | 1.10 (1.753) |  |  | 0.54 (0.923)
  Lymphocytes, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Lymphocytes, 48 hours | 5.18 (4.754) | 5.35 (5.907) | 4.39 (4.019) |
  Lymphocytes, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Lymphocytes, 72 hours | 5.15 (3.363) |  |  | 2.85 (7.766)
  Monocytes, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Monocytes, 48 hours | -0.13 (0.677) | 0.01 (1.093) | -0.12 (0.920) |
  Monocytes, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Monocytes, 72 hours | -0.18 (0.652) |  |  | 0.16 (1.249)
  Total neutrophils, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Total neutrophils, 48 hours | -6.56 (5.347) | -6.40 (7.071) | -5.10 (4.611) |
  Total neutrophils, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Total neutrophils, 72 hours | -6.20 (3.946) |  |  | -3.57 (9.212)

14. Primary Outcome: Change From Baseline in Hematology Parameter Hemoglobin for Part 1
Description: Blood samples were collected for the assessment of hematology parameter namely hemoglobin for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams/liter
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Grams/liter
  Hemoglobin, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Hemoglobin, 48 hours | 3.7 (4.66) | 4.8 (4.24) | 5.5 (5.05) |
  Hemoglobin, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Hemoglobin, 72 hours | 8.8 (5.23) |  |  | 5.0 (5.53)

15. Primary Outcome: Change From Baseline in Hematology Parameter Hematocrit for Part 1
Description: Blood samples were collected for the assessment of hematology parameter namely hematocrit for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Proportion of red blood cells in blood
  Hematocrit, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Hematocrit, 48 hours | 0.0188 (0.01542) | 0.0177 (0.01293) | 0.0238 (0.01599) |
  Hematocrit, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Hematocrit, 72 hours | 0.0255 (0.01472) |  |  | 0.0121 (0.01700)

16. Primary Outcome: Change From Baseline in Hematology Parameter Mean Corpuscle Hemoglobin for Part 1
Description: Blood samples were collected for the assessment of hematology parameter namely mean corpuscle hemoglobin for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Picograms
  Mean corpuscle hemoglobin, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Mean corpuscle hemoglobin, 48 hours | -0.32 (0.376) | -0.10 (0.429) | -0.14 (0.306) |
  Mean corpuscle hemoglobin, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Mean corpuscle hemoglobin, 72 hours | 0.22 (0.479) |  |  | 0.25 (0.362)

17. Primary Outcome: Change From Baseline in Hematology Parameter Mean Corpuscle Volume for Part 1
Description: Blood samples were collected for the assessment of hematology parameter namely mean corpuscle volume for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Femtoliters
  Mean corpuscle volume, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Mean corpuscle volume, 48 hours | 0.7 (0.78) | 0.3 (0.65) | 1.3 (0.87) |
  Mean corpuscle volume, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Mean corpuscle volume, 72 hours | 0.2 (0.75) |  |  | 0.2 (0.75)

18. Primary Outcome: Change From Baseline in Hematology Parameters Platelet Count and White Blood Cell Count for Part 1
Description: Blood samples were collected for the assessment of hematology parameters namely platelet count and white blood cell count for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga cells/liter
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Giga cells/liter
  Platelet count, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Platelet count, 48 hours | 3.7 (14.59) | 1.4 (12.55) | 0.5 (15.95) |
  Platelet count, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Platelet count, 72 hours | 14.5 (11.33) |  |  | 2.3 (10.53)
  White blood cell count,48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  White blood cell count,48 hours | -0.54 (0.489) | -0.48 (0.956) | -0.67 (0.947) |
  White blood cell count,72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  White blood cell count,72 hours | -0.32 (0.471) |  |  | -0.75 (1.258)

19. Primary Outcome: Change From Baseline in Hematology Parameters Red Blood Count and Reticulocyte Count for Part 1
Description: Blood samples were collected for the assessment of hematology parameters namely red blood count and reticulocyte count for Part 1. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Trillion cells/liter
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Trillion cells/liter
  Red blood cell count, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Red blood cell count, 48 hours | 0.165 (0.1650) | 0.164 (0.1385) | 0.197 (0.1797) |
  Red blood cell count, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Red blood cell count, 72 hours | 0.252 (0.1609) |  |  | 0.120 (0.1680)
  Reticulocyte count, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Reticulocyte count, 48 hours | 0.0127 (0.01512) | 0.0038 (0.01765) | -0.0009 (0.01929) |
  Reticulocyte count, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Reticulocyte count, 72 hours | -0.0023 (0.01646) |  |  | -0.0037 (0.01780)

20. Primary Outcome: Change From Baseline in Hematology Parameters Basophils, Eosinophils, Lymphocytes, Monocytes and Total Neutrophils for Part 2
Description: Blood samples were collected for the assessment of hematology parameters namely basophils, eosinophils, leukocytes, lymphocytes, monocytes, total neutrophils and platelets for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Percentage of cells
  Basophils, 48 hours | -0.00 (0.250) | 0.09 (0.120)
  Eosinophils, 48 hours | 0.44 (1.082) | 0.67 (0.960)
  Lymphocytes, 48 hours | 3.58 (7.821) | 4.53 (5.248)
  Monocytes, 48 hours | -0.04 (0.873) | -0.63 (0.936)
  Total neutrophils, 48 hours | -3.97 (9.311) | -4.66 (6.035)

21. Primary Outcome: Change From Baseline in Hematology Parameter Hemoglobin for Part 2
Description: Blood samples were collected for the assessment of hematology parameter namely hemoglobin for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams/liter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Grams/liter | 9.4 (3.92) | 8.9 (4.51)

22. Primary Outcome: Change From Baseline in Hematology Parameter Hematocrit for Part 2
Description: Blood samples were collected for the assessment of hematology parameter namely hematocrit for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Proportion of red blood cells in blood | 0.0304 (0.01286) | 0.0268 (0.01303)

23. Primary Outcome: Change From Baseline in Hematology Parameter Mean Corpuscle Hemoglobin for Part 2
Description: Blood samples were collected for the assessment of hematology parameter namely mean corpuscle hemoglobin for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Picograms | -0.12 (0.312) | 0.20 (0.268)

24. Primary Outcome: Change From Baseline in Hematology Parameter Mean Corpuscle Volume for Part 2
Description: Blood samples were collected for the assessment of hematology parameter namely mean corpuscle volume for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Femtoliters | 0.4 (0.96) | 0.6 (0.89)

25. Primary Outcome: Change From Baseline in Hematology Parameters Platelet Count and White Blood Cell Count for Part 2
Description: Blood samples were collected for the assessment of hematology parameters namely platelet count and white blood cell count for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga cells/liter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Giga cells/liter
  Platelet count, 48 hours | 7.4 (15.32) | 13.1 (12.45)
  White blood cell count,48 hours | 12.45 (0.995) | -0.36 (0.734)

26. Primary Outcome: Change From Baseline in Hematology Parameters Red Blood Count and Reticulocyte Count for Part 2
Description: Blood samples were collected for the assessment of hematology parameters namely red blood count and reticulocyte count for Part 2. Baseline was defined as assessments performed on Day -1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Trillion cells/liter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Trillion cells/liter
  Red blood cell count, 48 hours | 0.318 (0.1462) | 0.255 (0.1590)
  Reticulocyte count, 48 hours | -0.0018 (0.01203) | 0.0097 (0.01526)

27. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick Method for Part 1
Description: Urinalysis parameters assessed were urine bilirubin, urine occult blood, urine glucose, urine ketones, urine protein and urine urobilinogen. In this dipstick test, the level of bilirubin, occult blood, glucose, ketones, urine protein and urobilinogen in urine samples was recorded as negative, trace and +. Urine samples were collected for the measurement of urinalysis parameters by dipstick method up to 72 hours in Part 1. Only categories with significant values have been presented.
Time Frame: Up to 72 hours in Part 1
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Participants
  Urine occult blood, Trace, 48 hours | 1 | 1 | 0 | 0
  Urine occult blood, + , 48 hours | 0 | 1 | 1 | 0
  Urine occult blood, Trace, 72 hours | 1 | 0 | 0 | 0
  Urine occult blood, + , 72 hours | 1 | 0 | 0 | 0
  Urine protein, Trace, 48 hours | 0 | 1 | 1 | 0
  Urine protein, Trace, 72 hours | 1 | 0 | 0 | 0
  Urine urobilinogen, Trace, 48 hours | 12 | 12 | 12 | 0
  Urine urobilinogen, Trace, 72 hours | 6 | 0 | 0 | 11

28. Primary Outcome: Urine Potential of Hydrogen (pH) Analysis by Dipstick Method for Part 1
Description: Urinary pH measurement is a routine part of urinalysis. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Urine samples were collected for the measurement of urine pH by method up to 72 hours in Part 1. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
pH
  Urine pH, 48 hours: number analyzed (Participants) | 12 | 12 | 12 | 0
  Urine pH, 48 hours | 6.42 (0.634) | 6.17 (0.389) | 6.42 (0.469) |
  Urine pH, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Urine pH, 72 hours | 6.08 (0.492) |  |  | 6.36 (0.636)

29. Primary Outcome: Urine Specific Gravity Analysis by Dipstick Method for Part 1
Description: Urinary specific gravity measurement is a routine part of urinalysis. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Urine samples were collected for the measurement of urine specific gravity by dipstick method up to 72 hours in Part 1. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles). Density is the mass per unit volume and has units (such as g/cm^3), however, the specific gravity is a ratio so it has no unit.
Time Frame: Up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Ratio | 1.0167 (0.00753) | NA (NA) — NA indicates no sample was obtained per protocol for GSK1325756H 10 mg (fed) and GSK1325756H 50 mg (fed) at 72 hours post dose | NA (NA) — NA indicates no sample was obtained per protocol for GSK1325756H 10 mg (fed) and GSK1325756H 50 mg (fed) at 72 hours post dose | 1.0150 (0.00224)

30. Primary Outcome: Number of Participants With Abnormal Values on Urinalysis by Dipstick Method for Part 2
Description: Urinalysis parameters assessed were urine bilirubin, urine occult blood, urine glucose, urine ketones, urine protein and urine urobilinogen. In this dipstick test, the level of bilirubin, occult blood, glucose, ketones, urine protein and urobilinogen in urine samples was recorded as negative, trace and +. Urine samples were collected for the measurement of urinalysis parameters by dipstick method up to 48 hours in Part 2. Only categories with significant values have been presented.
Time Frame: Up to 48 hours in Part 2
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Participants
  Urine occult blood, Trace, 48 hours | 1 | 0
  Urine glucose, Trace , 48 hours | 1 | 0
  Urine protein, Trace, 48 hours | 0 | 2
  Urine urobilinogen, Trace, 48 hours | 15 | 15
  Urine urobilinogen, +, 48 hours | 1 | 1

31. Primary Outcome: Urine pH Analysis by Dipstick Method for Part 2
Description: Urinary pH measurement is a routine part of urinalysis. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Urine samples were collected for the measurement of urine pH by dipstick method up to 48 hours in Part 2.
Time Frame: Up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
pH | 6.66 (0.724) | 6.47 (0.718)

32. Primary Outcome: Urine Specific Gravity Analysis by Dipstick Method for Part 2
Description: Urinary specific gravity measurement is a routine part of urinalysis. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Urine samples were collected for the measurement of urine specific gravity by dipstick method up to 48 hours in Part 2. Density is the mass per unit volume and has units (such as g/cm^3), however, the specific gravity is a ratio so it has no unit.
Time Frame: Up to 72 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Ratio | 1.0153 (0.00618) | 1.0159 (0.00712)

33. Primary Outcome: Change From Baseline in Vital Sign Parameters Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) for Part 1
Description: Vital sign measurements included SBP and DBP at Baseline and up to 72 hours in Part 1. SBP and DBP measurements were preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions and were measured in a supine position after 5 minutes rest. Baseline was defined as pre-dose assessments performed on Day 1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Millimeters of mercury
  SBP, 4 hours | -4.8 (10.44) | -9.6 (9.21) | -4.2 (6.59) | -0.3 (7.02)
  SBP, 24 hours | 1.7 (7.95) | 0.5 (13.61) | 1.7 (6.87) | 4.5 (13.55)
  SBP, 48 hours | 4.5 (7.06) | 7.0 (10.76) | 5.9 (11.66) | 2.0 (10.47)
  SBP, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  SBP, 72 hours | -0.8 (8.06) |  |  | 4.8 (12.18)
  DBP, 4 hours | -3.6 (5.89) | -2.8 (3.33) | -2.2 (4.93) | -1.1 (5.36)
  DBP, 24 hours | 0.8 (4.94) | 4.5 (4.58) | 0.8 (6.40) | 1.0 (6.32)
  DBP, 48 hours | 2.0 (6.24) | 4.7 (6.07) | 2.1 (4.44) | 2.5 (6.12)
  DBP, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  DBP, 72 hours | 3.8 (4.12) |  |  | 1.8 (7.69)

34. Primary Outcome: Change From Baseline in Vital Sign Parameter Heart Rate for Part 1
Description: Vital sign measurements included heart rate at Baseline and up to 72 hours in Part 1. Heart rate measurements were preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions and were measured in a supine position after 5 minutes rest. Baseline was defined as pre-dose assessments performed on Day 1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Beats per minute
  Heart rate, 4 hours | -3.1 (3.92) | -3.2 (8.24) | -3.7 (6.17) | -2.9 (2.95)
  Heart rate, 24 hours | -3.0 (4.67) | -7.5 (9.23) | -3.8 (4.97) | -2.2 (4.07)
  Heart rate, 48 hours | -1.5 (3.09) | 1.2 (7.51) | -2.3 (6.59) | -2.7 (4.31)
  Heart rate, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Heart rate, 72 hours | -1.0 (4.98) |  |  | -1.0 (5.14)

35. Primary Outcome: Change From Baseline in Vital Sign Parameter Temperature for Part 1
Description: Vital sign measurements included temperature at Baseline and up to 72 hours in Part 1. Temperature measurements were preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions and were measured in a supine position after 5 minutes rest. Baseline was defined as pre-dose assessments performed on Day 1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Degree Celsius
  Temperature, 4 hours | 0.11 (0.363) | 0.07 (0.400) | 0.27 (0.393) | 0.14 (0.495)
  Temperature 24 hours | -0.08 (0.269) | 0.01 (0.375) | 0.06 (0.394) | 0.05 (0.321)
  Temperature, 48 hours | 0.02 (0.362) | -0.02 (0.364) | 0.01 (0.387) | 0.12 (0.460)
  Temperature, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Temperature, 72 hours | 0.00 (0.179) |  |  | 0.17 (0.272)

36. Primary Outcome: Change From Baseline in Vital Sign Parameters SBP and DBP for Part 2
Description: Vital sign measurements included SBP and DBP at Baseline and up to 72 hours in Part 2. SBP and DBP measurements were preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions and were measured in a supine position after 5 minutes rest. Baseline was defined as pre-dose assessments performed on Day 1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Millimeters of mercury
  SBP, 4 hours | -1.5 (11.70) | -2.5 (12.46)
  SBP, 24 hours | -2.8 (12.13) | -3.5 (11.64)
  SBP, 48 hours | -1.9 (10.22) | -0.2 (14.47)
  DBP, 4 hours | -0.8 (6.19) | -0.3 (6.63)
  DBP, 24 hours | -0.7 (6.66) | -0.6 (6.15)
  DBP, 48 hours | 0.1 (3.80) | 0.8 (6.31)

37. Primary Outcome: Change From Baseline in Vital Sign Parameter Heart Rate for Part 2
Description: Vital sign measurements included heart rate at Baseline and up to 72 hours in Part 2. Heart rate measurements were preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions and were measured in a supine position after 5 minutes rest. Baseline was defined as pre-dose assessments performed on Day 1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Beats per minute
  Heart rate, 4 hours | -2.4 (4.69) | -1.8 (5.14)
  Heart rate, 24 hours | 1.3 (5.46) | -0.1 (3.89)
  Heart rate, 48 hours | 0.5 (3.83) | 0.5 (4.07)

38. Primary Outcome: Change From Baseline in Vital Sign Parameter Temperature for Part 2
Description: Vital sign measurements included temperature at Baseline and up to 72 hours in Part 2. Temperature measurements were preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions and were measured in a supine position after 5 minutes rest. Baseline was defined as pre-dose assessments performed on Day 1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Degree Celsius
  Temperature, 4 hours | 0.06 (0.236) | 0.21 (0.340)
  Temperature 24 hours | 0.04 (0.250) | 0.10 (0.316)
  Temperature, 48 hours | 0.10 (0.228) | 0.10 (0.312)

39. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters PR Interval, QRS Duration, Uncorrected QT Interval and Corrected QT Frederica's Correction) Interval
Description: Single 12-lead ECG's were obtained from Baseline and up to 72 hours in Part 1 using an ECG machine that automatically calculated the heart rate and measured PR Interval, QRS Duration, Uncorrected QT interval and Corrected QT (Fridericia's correction) interval. Baseline was defined as pre-dose assessments performed on Day 1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value. Only those participants with data available at the specified time were analyzed (represented by n=x in the category titles).
Time Frame: Baseline and up to 72 hours in Part 1
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 18 | 12 | 12 | 11
Milliseconds
  PR Interval, 4 hours | -0.9 (11.65) | 0.7 (5.28) | 1.3 (4.29) | 0.5 (3.70)
  PR Interval 24 hours | 2.3 (5.63) | 3.0 (7.56) | 4.3 (6.20) | 3.6 (5.57)
  PR Interval, 48 hours | 5.6 (9.22) | -0.8 (8.50) | 5.7 (9.18) | 5.8 (6.84)
  PR Interval, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  PR Interval, 72 hours | 6.7 (11.57) |  |  | 6.0 (6.26)
  QRS duration, 4 hours | -0.4 (2.12) | -0.3 (2.39) | -0.2 (1.59) | -0.2 (3.03)
  QRS duration, 24 hours | 0.4 (1.89) | 0.7 (1.97) | 0.7 (1.56) | 0.4 (1.75)
  QRS duration, 48 hours | 1.0 (1.97) | 2.8 (1.99) | 1.7 (1.87) | 0.5 (2.02)
  QRS duration, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  QRS duration, 72 hours | 1.7 (2.34) |  |  | 0.9 (2.74)
  Uncorrected QT Interval, 4 hours | -1.7 (10.98) | -4.2 (15.90) | -4.0 (10.23) | -2.9 (11.08)
  Uncorrected QT Interval, 24 hours | -1.8 (10.74) | 6.8 (15.69) | -1.0 (9.82) | -1.5 (11.70)
  Uncorrected QT Interval, 48 hours | -4.4 (8.69) | -6.8 (12.52) | -1.5 (11.48) | -0.2 (14.76)
  Uncorrected QT Interval, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Uncorrected QT Interval, 72 hours | -8.3 (13.29) |  |  | -4.5 (14.54)
  Corrected QT Interval, 4 hours | -9.7 (5.32) | -11.3 (5.14) | -10.8 (7.16) | -8.1 (5.36)
  Corrected QT Interval, 24 hours | -7.6 (6.39) | -8.3 (7.75) | -9.5 (4.83) | -6.5 (6.02)
  Corrected QT Interval, 48 hours | -8.7 (6.45) | -5.9 (7.44) | -10.7 (6.51) | -6.9 (9.59)
  Corrected QT Interval,, 72 hours: number analyzed (Participants) | 6 | 0 | 0 | 11
  Corrected QT Interval,, 72 hours | -10.3 (3.27) |  |  | -7.6 (7.10)

40. Primary Outcome: Change From Baseline in Electrocardiogram Parameters PR Interval, QRS Duration, Uncorrected QT Interval and Corrected QT (Frederica's Correction) Interval for Part 2
Description: Single 12-lead ECG's were obtained from Baseline and up to 72 hours in Part 2 using an ECG machine that automatically calculated the heart rate and measured PR Interval, QRS Duration, Uncorrected QT interval and Corrected QT (Frederica's correction) interval. Baseline was defined as pre-dose assessments performed on Day 1. Change from Baseline was calculated by subtracting the post-dose-visit value from the Baseline value.
Time Frame: Baseline and up to 48 hours in Part 2
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Milliseconds
  PR Interval, 4 hours | -1.5 (5.59) | -0.6 (4.18)
  PR Interval 24 hours | -2.5 (7.50) | 1.3 (4.37)
  PR Interval, 48 hours | 1.5 (8.84) | 4.1 (6.13)
  QRS duration, 4 hours | -0.6 (2.28) | -1.3 (4.12)
  QRS duration, 24 hours | -1.0 (2.19) | -1.8 (5.00)
  QRS duration, 48 hours | -0.6 (2.50) | -0.9 (4.26)
  Uncorrected QT Interval, 4 hours | 3.1 (12.31) | 6.4 (10.02)
  Uncorrected QT Interval, 24 hours | -10.0 (15.85) | -3.9 (13.83)
  Uncorrected QT Interval, 48 hours | -6.4 (11.25) | -9.5 (17.84)
  Corrected QT Interval, 4 hours | -3.1 (6.55) | 3.1 (7.20)
  Corrected QT Interval, 24 hours | -6.1 (6.73) | -3.8 (7.38)
  Corrected QT Interval, 48 hours | -5.7 (5.58) | -7.3 (8.69)

41. Primary Outcome: Blood Concentration of GSK1325756 in Part 1
Description: Whole blood samples of approximately 1 milliliters were collected for measurement of blood concentrations of GSK1325756 at pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in all 3 periods; 60 and 72 hours post-dose in period-3 of part 1. Data has been presented for blood concentrations of GSK1325756 in fed state. Pharmacokinetic (PK) population was defined as participants who were administered at least one dose of study treatment and who had PK sample taken and analyzed. NA indicates standard deviation could not be calculated due to high proportion of non-quantifiable [NQ] values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation and no sample was obtained per protocol for 60 and 72 hours.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in all 3 periods; 60 and 72 hours post-dose in period-3 of Part 1
Population: PK Population
Measure: Mean (Standard Deviation); unit: Nanograms/milliliter
Arm/Group | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 12 | 12 | 11
Nanograms/milliliter
  Blood concentration, Pre-dose | 0.000 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation. | 0.000 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation. | 0.000 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation.
  Blood concentration, 0.25 hours | 1.425 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation. | 9.289 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation. | 32.318 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation.
  Blood concentration, 0.5 hours | 24.350 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation. | 151.658 (196.5556) | 201.782 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation.
  Blood concentration, 0.75 hours | 59.951 (67.9706) | 373.193 (376.8749) | 426.032 (611.1420)
  Blood concentration, 1 hour | 94.150 (86.0423) | 455.042 (350.7416) | 634.955 (767.2316)
  Blood concentration,, 2 hours | 153.395 (100.0463) | 971.417 (598.1981) | 1285.524 (1017.193)
  Blood concentration, 3 hours | 154.733 (67.6734) | 950.852 (443.1637) | 1235.273 (740.0601)
  Blood concentration, 4 hours | 177.417 (47.6187) | 966.658 (395.2375) | 1498.000 (607.8816)
  Blood concentration, 6 hours | 126.817 (37.7057) | 639.667 (251.0068) | 1418.545 (497.2105)
  Blood concentration, 8 hours | 76.567 (25.8472) | 386.667 (153.4840) | 735.700 (234.1135)
  Blood concentration, 10 hours | 55.358 (16.1098) | 295.250 (96.3848) | 620.636 (217.5446)
  Blood concentration,12 hours | 39.742 (10.1591) | 204.192 (70.3804) | 411.091 (143.5280)
  Blood concentration, 24 hours | 16.363 (4.9104) | 77.342 (37.3054) | 160.982 (61.3081)
  Blood concentration, 48 hours | 3.423 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation. | 24.387 (13.2219) | 43.282 (17.8091)
  Blood concentration, 60 hours | NA (NA) — NA indicates no sample obtained per protocol. | NA (NA) — NA indicates no sample obtained per protocol. | 19.087 (11.6452)
  Blood concentration, 72 hours | NA (NA) — NA indicates no sample obtained per protocol. | NA (NA) — NA indicates no sample obtained per protocol. | 18.403 (12.5176)

42. Primary Outcome: Blood Concentration of GSK1325756 in Part 2
Description: Whole blood samples of approximately 1 milliliters were collected for measurement of blood concentrations of GSK1325756 at Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose in part 1. Data has been presented for blood concentrations of GSK1325756 in fasted and fed state. NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose in Part 2
Population: PK Population
Measure: Mean (Standard Deviation); unit: Nanograms/milliliter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Nanograms/milliliter
  Blood concentration, Pre-dose | 0.000 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation. | 0.000 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation.
  Blood concentration, 0.25 hours | 23.888 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation. | 434.557 (551.7663)
  Blood concentration, 0.5 hours | 248.749 (NA) — NA indicates standard deviation could not be calculated due to high proportion of NQ values (more than 30% of values were imputed i.e., NQ assigned zero concentration) which affected the standard deviation. | 2233.813 (1476.075)
  Blood concentration, 0.75 hours | 363.644 (745.3481) | 3599.500 (1240.578)
  Blood concentration, 1 hour | 470.700 (711.2266) | 4210.625 (1361.315)
  Blood concentration, 2 hours | 1039.688 (638.7844) | 3176.000 (691.7762)
  Blood concentration, 3 hours | 1499.250 (657.7378) | 2156.250 (521.9307)
  Blood concentration, 4 hours | 1682.667 (478.1134) | 1960.625 (402.0194)
  Blood concentration, 6 hours | 774.938 (305.5721) | 640.500 (140.6840)
  Blood concentration, 8 hours | 463.750 (143.7101) | 410.625 (105.4564)
  Blood concentration, 10 hours | 364.438 (117.3348) | 350.813 (112.8440)
  Blood concentration,12 hours | 244.938 (76.6059) | 254.188 (68.8847)
  Blood concentration, 24 hours | 111.163 (43.6251) | 118.888 (53.3676)
  Blood concentration, 48 hours | 40.568 (61.6334) | 29.918 (32.5396)

43. Primary Outcome: Maximum Observed Concentration (Cmax) of GSK1325756H for Part 1
Description: Blood samples were collected at the indicated time points after administration of study treatment to investigate the PK profile of GSK1325756H in fasted state. PK parameters were calculated by standard non-compartmental analysis using Phoenix WinNonlin Version 6.4 or higher based on actual sampling times.
Time Frame: as for outcome 41
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter
Groups:
- Part 1:GSK1325756H 50 mg (Fed): Participants received GSK1325756H 50 mg tablets via the oral route with food (fed state) and 240 milliliters of water in Part 1.
Arm/Group | Part 1: GSK1325756H 10 mg (Fed) | Part 1:GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 12 | 12 | 11
Nanograms/milliliter | 217.082 (17.8) | 1219.883 (37.3) | 1924.864 (39.6)

44. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to t (AUC [0-t]) of GSK1325756H for Part 1
Description: as for outcome 43
Time Frame: as for outcome 41
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 12 | 12 | 11
Hours*nanograms/milliliter | 1622.2891 (21.7) | 8872.6074 (30.2) | 16681.8331 (25.2)

45. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC [0-inf]) of GSK1325756H for Part 1
Description: as for outcome 43
Time Frame: as for outcome 41
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 12 | 12 | 11
Hours*nanograms/milliliter | 1779.0163 (18.8) | 9253.2108 (31.3) | 17072.6642 (24.4)

46. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 Hours (AUC [0-24]) of GSK1325756H for Part 1
Description: as for outcome 43
Time Frame: as for outcome 41
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 12 | 12 | 11
Hours*nanograms/milliliter | 1500.0109 (14.7) | 7831.8861 (29.9) | 14000.5473 (27.1)

47. Primary Outcome: Time to Maximum Observed Concentration (Tmax) of GSK1325756H for Part 1
Description: as for outcome 43
Time Frame: as for outcome 41
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 12 | 12 | 11
Hours | 3.50000 [2.0000 to 6.0000] | 3.00000 [2.0000 to 6.0000] | 4.00000 [2.0000 to 6.0000]

48. Primary Outcome: Terminal Half-life (t1/2) of GSK1325756H for Part 1
Description: Blood samples were collected at the indicated time points after administration of study treatment to investigate the PK profile of GSK1325756 in fasted state. PK parameters were calculated by standard non-compartmental analysis using Phoenix WinNonlin Version 6.4 or higher based on actual sampling times.
Time Frame: as for outcome 41
Population: PK Population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 12 | 12 | 11
Hours | 10.53043 (2.938579) | 11.17318 (2.284423) | 13.15755 (4.540486)

49. Primary Outcome: Lag Time Before Observable Concentration (Tlag) of GSK1325756H for Part 1
Description: as for outcome 48
Time Frame: as for outcome 41
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 12 | 12 | 11
Hours | 0.37500 [0.0000 to 1.0000] | 0.25000 [0.0000 to 2.0000] | 0.25000 [0.0000 to 1.0000]

50. Primary Outcome: Time to Last Quantifiable Concentration (Tlast) of the Blood Concentration of GSK1325756H for Part 1
Description: as for outcome 43
Time Frame: as for outcome 41
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed)
Number analyzed (Participants) | 12 | 12 | 11
Hours | 36.00000 [24.0000 to 48.0000] | 48.00000 [48.0000 to 48.0000] | 72.00000 [48.0000 to 72.0000]

51. Primary Outcome: Cmax of GSK1325756H for Part 2
Description: as for outcome 43
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Nanograms/milliliter | 1818.544 (32.5) | 4146.886 (34.5)

52. Primary Outcome: AUC (0-t) of GSK1325756H for Part 2
Description: as for outcome 43
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Hours*nanograms/milliliter | 11880.9038 (28.9) | 18303.0441 (22.1)

53. Primary Outcome: AUC (0-inf) of GSK1325756H for Part 2
Description: Blood samples were collected at the indicated time points after administration of study treatment to investigate the PK profile of GSK1325756H in fasted state. PK parameters were calculated by standard non-compartmental analysis using Phoenix WinNonlin Version 6.4 or higher based on actual sampling times. Only those participants with data available at the indicated time points were analyzed.
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 15 | 16
Hours*nanograms/milliliter | 12143.8862 (28.8) | 18910.7975 (24.2)

54. Primary Outcome: AUC (0-24) of GSK1325756H for Part 2
Description: as for outcome 43
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose in Part 2
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Hours*nanograms/milliliter | 10433.9293 (25.8) | 16856.0664 (21.2)

55. Primary Outcome: Tmax of GSK1325756H for Part 2
Description: as for outcome 43
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose in Part 2
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Hours | 3.00000 [0.5000 to 6.0000] | 1.00000 [0.5000 to 3.0000]

56. Primary Outcome: t1/2 of GSK1325756H for Part 2
Description: as for outcome 53
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose in Part 2
Population: PK Population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 15 | 16
Hours | 10.75500 (2.928804) | 11.09246 (5.259109)

57. Primary Outcome: Tlag of GSK1325756H for Part 2
Description: as for outcome 43
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose in Part 2
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Hours | 0.25000 [0.0000 to 1.0000] | 0.00000 [0.00000 to 0.00000]

58. Primary Outcome: Tlast of the Blood Concentration of GSK1325756H for Part 2
Description: as for outcome 43
Time Frame: Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 post-dose in Part 2
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
Number analyzed (Participants) | 16 | 16
Hours | 48.00000 [24.0000 to 48.0000] | 48.00000 [48.0000 to 48.0000]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the Day -1 up to follow-up ( 32 days for Part 1 and up to 21 days for Part 2)
Description: Safety Population was used for analysis of AE and SAE's.
Groups:
- Part 2: GSK1325756H 50 mg (Fasted): Participants received GSK1325756H 50 mg tablets via the oral route without food (fasted state) and 240 mililiters of water in Part 2.
Arm/Group | Part 1: Placebo (Fed) | Part 1: GSK1325756H 10 mg (Fed) | Part 1: GSK1325756H 50 mg (Fed) | Part 1: GSK1325756H 100 mg (Fed) | Part 2: GSK1325756H 50 mg (Fed) | Part 2: GSK1325756H 50 mg (Fasted)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/12 | 0/12 | 0/11 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/12 | 0/12 | 0/11 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/18 | 0/12 | 0/12 | 1/11 | 1/16 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (Fed) (N=18) | Part 1: GSK1325756H 10 mg (Fed) (N=12) | Part 1: GSK1325756H 50 mg (Fed) (N=12) | Part 1: GSK1325756H 100 mg (Fed) (N=11) | Part 2: GSK1325756H 50 mg (Fed) (N=16) | Part 2: GSK1325756H 50 mg (Fasted) (N=16)
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT03136380/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03136380/SAP_001.pdf